CLINICAL TRIAL: NCT03778541
Title: Hypofractionated Radiotherapy With Concurrent Temozolomide for Large Brain Metastases: a Multi-center Randomized Phase III Trial
Brief Title: HFSRT With Concurrent TMZ for Large BMs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBM-RCT
Record Dates: First submitted 2018-12-09; First posted 2018-12-19 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Brain Metastases; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide; Radiation Dose Hypofractionation

STUDY DESIGN:
Intervention Model Description: patients were randomized to 2 parallel groups, namely the concurrent chemoradiotherapy group and radiotherapy alone group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRT group (Experimental): patients with brain metastases of more than 6 cc and treated with fractionated stereotactic radiotherapy plus concomitant Temozolomide.
  Interventions: Drug: Temozolomide; Radiation: hypofractionated radiotherapy
- RT group (Active Comparator): patients with brain metastases of more than 6 cc and treated with fractionated stereotactic radiotherapy alone.
  Interventions: Radiation: hypofractionated radiotherapy

INTERVENTIONS:
Drug: Temozolomide — 75mg/m2/d concurrent with radiotherapy, taken for at least 20 days.
  Arms: CRT group
Radiation: hypofractionated radiotherapy — the regular radiation dose prescription is 52 Gy in 13 fractions or 52.5 Gy in 15 fractions.

SUMMARY:
A multi-center randomized phase III trial was conducted to investigate the feasibility and safety of adding temozolomide to hypofractionated stereotactic radiotherapy for large brain metastases.

DETAILED DESCRIPTION:
A previous single arm phase II trial and propensity- matched study of our institution have shown that HFSRT combined with concurrent TMZ was safe and efficient for patients with BMs of ≥ 6cc in volume. The 1-year local control, intracranial progression free survival, progression free survival and overall survival rates were better than HFSRT alone group. Thus, the investigator conducted this randomized phase III trial to broad the sample size and verify our previous results. To finish the study in time, the investigator designed a multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytological diagnosis of primary tumor and conformed brain metastases by enhanced MRI or CT;
* the number of BMs ≤ 3
* the tumor volume ≥6cc, or maximum diameter of BMs≥ 3cm;
* Karnofsky performance score (KPS)≥60, or KPS≥40 but simply caused by BMs;
* Age: 18-75 years old;
* Adequate function of major organs, and blood test reached the following level: WBC≥4.0x109/L, NEU≥1.5x109/L Hemoglobin≥110 g/L, Platelets≥100 x109/L; Liver function test results<1.5 times the institutional upper limit of normal (ULN); BUN and Cr: within the normal range.

Exclusion Criteria:

* patient with other clinically significant diseases (e.g. myocardial infarction within the past 6 months, severe arrhythmia);
* unable or unwilling to comply with the study protocol;
* patient whose survival expectancy was less than 3 months;
* the large BM locates in brainstem;
* patient who anticipated in other clinical trials of brain metastases;
* the large lesions have been treated with SRT in other hospitals;
* pregnant patients or female patients whose HCG is positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-12-03 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
intracranial progression free survival (IPFS) rate | up to 2 years
  IPFS was defined as the interval from the beginning of radiation to any intracranial progression

SECONDARY OUTCOMES:
local control rate | up to 2 years
  the control rate of treated lesions
Brain metastasis-specific survival (BMSS) rate | up to 2 years
  BMSS was defined as the internal from the beginning of RT to death caused by BM
overall survival (OS) rate | up to 2 years
  OS was defined as the internal from the beginning of RT to death caused by any reason
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 and NRG/RTOG CNS toxicities criteria | acute toxicities: up to 3 months after RT; Late toxicities: up to 2 years after RT
  the toxicities caused by RT and (or) Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Dr, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No